CLINICAL TRIAL: NCT02899624
Title: Whole Exome Sequencing in Bicuspid Aortic Valve Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-09
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Bicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bicuspid aortic valve (BAV) (Experimental): patient with bicuspid aortic valve
  Interventions: Biological: Extra blood draw samples; Biological: additional tissue samples
- healthy subjects related patients with BAV (Active Comparator): healthy control, related to patient with bicuspid aortic valve, at the 1st, 2nd or 3rd degree
  Interventions: Biological: Extra blood draw samples
- Tricuspid aortic valve (TAV) (Active Comparator): patient with aortic stenosis on tricuspid valve
  Interventions: Biological: additional tissue samples

INTERVENTIONS:
Biological: Extra blood draw samples
  Arms: Bicuspid aortic valve (BAV); healthy subjects related patients with BAV
Biological: additional tissue samples
  Arms: Bicuspid aortic valve (BAV); Tricuspid aortic valve (TAV)

SUMMARY:
Bicuspid aortic valve (BAV), congenital anomaly present in 2% of the population, is defined by the presence of two sigmoid valves instead of three. It is conventionally associated with histological abnormalities of the wall of the ascending aorta, risk factors of aortic dystrophy observed in 50% of cases, and dissection. Long considered an accident of development, the discovery of mutations in the NOTCH1 gene in 2 families alternating BAV and aortic dystrophy suggests the existence of a genetic predisposition and a common genetic origin for these two pathologies.

Data on the genetic basis of the BAV are still limited, but the existence of a large phenotypic diversity suggests the involvement of other genes. The establishment of large collections of DNA will allow great advances in this field.

The purpose of this project is to confirm the existence of a genetic determinism at the origin of the BAV with or without dystrophy of non syndromic ascending aorta, identifying genetic defects associated with the presence of a BAV in a series of candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* bicuspid aortic valve, confirmed by transthoracic or transesophageal echocardiography
* With or without an aneurysm of the ascending thoracic aorta nonsyndromic

Exclusion Criteria:

* aortic syndromic pathology
* antecedent of acute articular rhumatism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
number of genetic abnormalities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No